CLINICAL TRIAL: NCT07266324
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2 Study to Assess Efficacy, Safety and Tolerability of BMB-101 Oral Solution for the Treatment of Patients With Prader-Willi Syndrome (PWS)
Brief Title: A 2-Part Study to Assess Efficacy, Safety and Tolerability of BMB-101 for the Treatment of Patients With Prader-Willi Syndrome.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bright Minds Biosciences Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BMB-101-201
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMB-101 (Experimental): Participants receive BMB-101 (10mg/mL liquid) orally
  Interventions: Drug: BMB-101
- Placebo (Placebo Comparator): Participants receiving matched placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMB-101 — Participants will receive weekly ascending oral doses of BMB-101(10 mg/mL) twice daily (BID) for 16 weeks.
  Doses will be based on weight (kg) and will initially start at 1.67 mg/kg. Doses may be titrated in 0.33 mg/kg increments based on tolerability up to a maximum dose of 2.0 mg/kg.
  Arms: BMB-101
Drug: Placebo — Matched Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the safety and effects of a new drug called BMB-101 in people with Prader-Willi Syndrome (PWS). This study is designed as a multi-centre, double-blind, randomized, placebo controlled 2-part study with a blinded main phase followed up an open label extension phase.

DETAILED DESCRIPTION:
This study is designed as a 2-part study:

Part 1 is designed as a randomized phase, lasting up to 16 weeks. There will be a 4-week screening period. Following the screening period, participants will be randomized in a 1:1 ratio to either BMB-101 or placebo. Participants will enter into a weekly ascending Maximum Tolerated Dose (MTD) titration phase of 4 weeks followed by a maintenance phase of 8 weeks. There will be 5 clinic visits and 4 telephone visits.

Part 2 is designed to follow after the completion of the maintenance phase in Part 1. Participants at the discretion of the Investigator may elect to continue into an unblinded, expandable open label phase to receive BMB-101.

Participants who do not elect to continue into the open label phase will be tapered from assigned study treatment over 4 weeks following completion of the maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be aged 18-65 years (both inclusive).
* Genetically confirmed diagnosis of Prader Willi Syndrome via standard DNA testing or other commonly approved methods.
* Willing and able to provide voluntary written informed consent, or have a Legally Authorized Representative who is able to provide consent.
* Moderate to severe hyperphagia as defined by a HQ-CT score ≥ 13 at time of randomization (Visit 3).
* If participant is receiving growth hormone, the subject must be on the same medication and stable dose for at least 90 days prior to Visit 1.
* Female participant of childbearing potential must have a negative urine pregnancy test at baseline. Participants of childbearing or child-fathering potential must be willing to use medically acceptable forms of birth control, which includes abstinence, while in this study and for 90 days after the last dose of study drug.
* Participant and/or caregiver has the ability to be compliant with study requirements, including visit schedule, diary completion and study drug accountability.
* If a caregiver assists in completion of questionnaires, the same caregiver is available to complete the questionnaires throughout the duration of the study.

Exclusion Criteria:

* Participant has used metabolic agents known to affect appetite within 3 months of Visit 1.
* Participant use of psychotropic medications including SSRIs/SNRIs, monoamine-oxidase inhibitors, tricyclic antidepressants, other serotonergic agonists or antagonists (antipsychotics), and other agents which have known Serotonin Syndrome risk (e.g. mirtazapine) within 1 month of Visit 1.
* Participant has implementation of new food restrictions or new environmental restrictions within 1 month of Visit 1.
* Participant has participated in an interventional clinical trial of any Prader-Willi Syndrome agent within 3 months of Visit 1 or any other investigational agent within 1 month of Visit 1.
* Participant has current or past history of cardiovascular or cerebrovascular disease, such as cardiac valvulopathy, pulmonary hypertension, myocardial infarction or stroke, or clinically significant structural cardiac abnormality.
* Participant has moderate or severe hepatic impairment. Asymptomatic participants with mild hepatic impairment (elevated liver enzymes < 3x upper limit of normal (ULN) and/or elevated bilirubin <2x ULN) may be entered into the study after review and approval by the Medical Monitor in conjunction with the sponsor, in consideration of comorbidities and concomitant medications.
* Participant has severe renal impairment (estimated glomerular filtration rate <30mL/min/1.73m2).
* Participant has clinically significant ECG abnormality such as QTcF >450 msec (males) or >470 msec (females).
* Participant has a history of drug or alcohol abuse within the last 12 months or a positive urine drug screen.
* A current C-SSRS score of 4 or 5 at Visit 1 or history of suicide attempt at any time during the past year.
* Participant has a clinically significant condition or has had clinically relevant symptoms or a clinically significant illness in the 4 weeks prior to Visit 1, other than PWS, that would negatively impact study participation, collection of study data, evaluation of study endpoints or pose a risk to the participant, in the opinion of the Investigator.
* Participant is pregnant (determined by a positive urine pregnancy test) or lactating female.
* Any condition that is thought to be a degenerative neurological disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hyperphagia Questionnaire for Clinical Trials scores over time in Prader-Willi Syndrome participants. | 16 weeks
  The Hyperphagia Questionnaire for Clinical Trials consists of 9 items; each rated on a scale from 0 (no symptoms) to 4 (severe symptoms). The total score ranges from 0 to 36, with higher scores indicating worse hyperphagia symptoms. A score of approximately 13 is associated with moderate to severe hyperphagia, and a score of 22 or greater is associated with severe hyperphagia.

SECONDARY OUTCOMES:
Change from Baseline in hyperphagia severity score as measured by the Caregiver Global Impression of Severity 7-point scale over time. | 16 weeks
  This scale is a single-item measure from 1 to 7, where higher scores indicate greater severity.
Change from Baseline in hyperphagia severity score as measured by the Clinician Global Impression of Severity 7-point scale over time. | 16 weeks
  This scale is a single-item measure from 1 to 7, where higher scores indicate greater severity.
Change from Baseline in severity of Prader-Willi Syndrome disease scores as measured by the Clinician Global Impression of Severity 7-point scale over time. | 16 weeks
  This scale is a single-item measure from 1 to 7, where higher scores indicate greater severity.
Change from Baseline in improvement of Prader-Willi Syndrome disease scores as measured by the Clinician Global Impression of Improvement 7-point scale over time. | 16 weeks
  This scale is a single-item measure from 1 to 7, where 1 indicates very much improved, and 7 indicates very much worse.
Change from Baseline in Prader-Willi Syndrome correlated behavioral issues such as symptoms measured by the Prader-Willi Syndrome Profile on a 3-point scale over time. | 16 weeks
  The Prader-Willi Syndrome Profile is a 57-item caregiver rated questionnaire that measures 52 Prader-Willi Syndrome specific behaviors on a 3-point scale (0-2), where 0=Not True, and 2=Often True. Higher scores indicate greater severity.

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Alfred Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No